CLINICAL TRIAL: NCT00754533
Title: Influence of Different Exercise Training Programs in Patients With Coronary Artery Disease on Cardiac and Respiratory Parameters
Brief Title: Continuous Versus Interval Training in Patients With Coronary Artery Disease: FRAXIO Study
Acronym: FRAXIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: SENGELEN Marie / Directrice des Affaires Médicales et de la Recherche Clinique, University Hospital, Limoges
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I08005
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2008-10

CONDITIONS: Acute Coronary Syndrome
Keywords: cardiac rehabilitation; coronary heart disease; interval training; continuous training; ventilatory threshold
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Continuous training
  Interventions: Other: Continuous versus interval training
- 2 (Other): Interval training
  Interventions: Other: Continuous versus interval training

INTERVENTIONS:
Other: Continuous versus interval training — Influence of different exercise training programs

SUMMARY:
The benefits of cardiac rehabilitation have been clearly demonstrated. In particular exercise training is recognized to be part of modern management after coronary artery disease. However methods of prescribing exercise-training programs and the exercise intensity are difficult to determine. The objective of this randomised clinical trial is to determine whether appropriate endurance exercise training improves the ventilatory threshold, the exercise tolerance and the quality of life in patients with coronary artery disease. Patients are randomized to continuous training or aerobic interval training respectively: 80%-versus maximal-workload at the ventilatory threshold. For each patient, the intensity of exercise training is determined by a first exercise test with gas analysis using parameters of sub maximal exercise capacity such as ventilatory threshold. Others parameters of functional capacity are also considered. Duration of the rehabilitation stage is between 7 to 10 weeks. Dyspnoea assessment at maximal intensity, quality of life measurement by SF36, drugs and events are reported. Maximal exercise tests with gas exchange measurements are performed after training program and at 6 months follow-up to compare the different cardio respiratory parameters in the two groups before and after exercise training and to evaluate the more effective endurance training program.

DETAILED DESCRIPTION:
* Outline of the training program: Duration of the rehabilitation course is 7 or 10 weeks, 2 or 3 training sessions a week, 21 sessions altogether. Each training session consist in cycling on an ergometer. In the interval training group, the training session alternates one minute at 100% workload at the ventilatory threshold and one minute active pause at 50% workload at the ventilatory threshold; total exercise time is 20 minutes. In continuous training, the training session lasts 20 minutes at 80% workload at the ventilatory threshold.
* Exercise testing: Exercise capacity is measured before and at the end of the exercise training program and at 6 month follow-up. A first exercise test with respiratory gas exchange is performed 2 weeks after hospitalization: this is the baseline exercise test. The protocol consists of 3-min warm up at a workload of 30 watts. At each stage, the workload is increased by 10 or 15 watts per min. Patients are instructed to maintain a speed of 55 to 65 rotations per min. Four exercise tests with gas analysis are programmed during cardiac rehabilitation: three maximal tests (before exercise training program to precise exercise intensity during the sessions, after training program to evaluate the primary end point and at 6 months) and one sub maximal exercise test during the tenth session to adjust the intensity of training exercises (this test is stopped when the ventilatory threshold is obtained).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient hospitalized at Limoges University Hospital, cardiology department, for acute coronary syndrome:

  * with or without ST segment elevation
  * with or without elevated troponin
  * with or without revascularization
* Patients stabilized with medication without rest myocardial ischemia
* Left ventricular ejection fraction >= 35% measured on echocardiography
* Patient who have signed and dated informed consent
* Patient who can do a maximal metabolic exercise test

Exclusion Criteria:

* Contraindication for exercise testing:

  * acute myocardial infraction < 5 days
  * unstable angina
  * left main coronary stenosis
  * uncontrolled cardiac arrhythmia
  * uncontrolled symptomatic heart failure
  * acute pulmonary embolism or phlebitis
  * acute myocarditis, pericarditis or endocarditis
  * patient's physical inability or refusal
  * left ventricular thrombus after acute myocardial infarction
  * pulmonary hypertension > 60 mmHg
  * uncontrolled arterial hypertension
* Age < 18 years
* Patient revascularized by coronary artery bypass grafting after acute coronary syndrome
* Chronic supraventricular arrhythmias
* Impossible physical exercise
* Patient who can't understand the protocol or who refused to give his consent
* Patient who already attended a training program over the last 6 months
* Patient with difficult follow-up
* Current participation in another study
* Patient under guardianship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is to compare the effect on ventilatory threshold before and after cardiac rehabilitation in the continuous training group versus interval training group | 6 month

SECONDARY OUTCOMES:
The secondary endpoint is to compare the effect on ventilatory threshold before and at 6 month after cardiac rehabilitation in the two groups | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Prisca DEMAISON, MD, Principal Investigator — University Hospital, Limoges
Locations (2):
- France (2):
  - Cardiology, Limoges
  - Explorations Fonctionnelles Physiologiques, Limoges